CLINICAL TRIAL: NCT05450809
Title: PeRfOrmance and ACcuracy of an artifiCial Intelligence Enhanced Smart Watch Single Lead ECG (PROCESS)
Brief Title: Performance and Accuracy of an AI Enhanced Smart Watch Single Lead ECG
Acronym: PROCESS
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Itzhak Zachi Attia, Principal Investigator, Mayo Clinic
Other Study IDs: 21-006770
Record Dates: First submitted 2022-07-05; First posted 2022-07-11 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Healthy
Keywords: electrocardiogram; wearable; artificial intellegence; Apple Watch

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Ambulatory, outpatient Mayo Clinic ECG lab patients: Patients who are undergoing routine clinical evaluation with a 12 lead ECG recording ordered at the Mayo Clinic ECG lab.

SUMMARY:
The purpose of this study is to show the artificial intelligence enhanced single-lead ECG Apple Watch has similar, robust performance comparable to an AI enhanced 12 lead ECG and AI enhanced single lead (LI) of a 12 lead ECG.

DETAILED DESCRIPTION:
1. Ambulatory patients undergoing ECG recording in the Mayo Clinic outpatient ECG lab will be asked to consent for this study.
2. Those who consent for the study will be asked to record a ECG using a single-lead watch-based (Apple Watch series 5) recording at a visit for a clinically scheduled 12 lead ECG recording.
3. This watch-based ECG data will be recorded and analyzed in comparison to the near-simultaneously recorded outpatient 12 Lead ECG

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and ≤ 89.
* Able to give verbal consent.
* Able to complete routine clinical 12 lead ECG tracing and single lead Apple Watch ECG tracing.

Exclusion Criteria:

* Individuals < 18 and > 89 years of age.
* Unable to given verbal consent.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ambulatory patients who are undergoing a clinically ordered electrocardiogram in the Mayo Clinic outpatient ECG lab.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2021-11-05 (Actual); Primary Completion 2022-11-02 (Actual); Study Completion 2022-11-02 (Actual)

PRIMARY OUTCOMES:
Comparison of 12 lead ECG features to single-lead watch-based ECG features | 12 months
  The ECG interval differences (in milliseconds) between 12 Lead and collected single-lead watch-based ECG for PR, QRS, QT intervals will be determined and compared for each patient.
Arrhythmia comparison of 12 lead ECG to single-lead watch-based ECG | 12 months
  A physician interpretation of patients' 12 lead ECG and single-lead watch-based ECG will be performed to determined underlying rhythm (i.e. sinus rhythm, atrial fibrillation etc) from each, and the results from these modalities will be compared.

SECONDARY OUTCOMES:
Arrhythmia classification by physician overread of single-lead watch-based ECG | 12 months
  A physician interpretation of the patient's single-lead watch-based ECG will occur as described in "Outcome 2." The results of this ECG interpretation (i.e. sinus rhythm, atrial fibrillation, or inconclusive) will be compared to the watch/app-based rhythm auto-classification for each recorded single-lead watch-based ECG.

OTHER OUTCOMES:
Artificial intelligence detection of heart failure by single-lead watch-based ECG | 12 months
  A previously developed AI algorithm to predict potential underlying cardiac pathology assess from 12 lead ECG via convolutional neural network will be adapted applied to the ECGs for patients who undergo single-lead watch-based ECG recording. This neural network uses PQRST complexes to yield a probability of heart failure which may not be readily apparent via manual review. Each recorded single-lead watch-based ECG will undergo evaluation by this neural network and will produce a probability of heart failure (0-100%) for each individual patient. This probability will be compared to the AI ECG result (probability 0-100%) from the patient's recently recorded 12 lead ECG which is routinely available for all patients with a recorded 12 lead ECG at our medical system.
Artificial intelligence detection of silent/paroxysmal atrial fibrillation by single-lead watch-based ECG | 12 months
  A previously developed AI algorithm to predict potential underlying cardiac pathology assess from 12 lead ECG via convolutional neural network will be adapted applied to the ECGs for patients who undergo single-lead watch-based ECG recording. This neural network uses PQRST complexes to yield a probability of silent/paroxysmal atrial fibrillation which may not be readily apparent via manual review. Each recorded single-lead watch-based ECG will undergo evaluation by this neural network and will produce a probability of silent/paroxysmal atrial fibrillation (0-100%) for each individual patient. This probability will be compared to the AI ECG result (probability 0-100%) from the patient's recently recorded 12 lead ECG which is routinely available for all patients with a recorded 12 lead ECG at our medical system.
Artificial intelligence detection of aortic stenosis by single-lead watch-based ECG | 12 months
  A previously developed AI algorithm to predict potential underlying cardiac pathology assess from 12 lead ECG via convolutional neural network will be adapted applied to the ECGs for patients who undergo single-lead watch-based ECG recording. This neural network uses PQRST complexes to yield a probability of aortic stenosis which may not be readily apparent via manual review. Each recorded single-lead watch-based ECG will undergo evaluation by this neural network and will produce a probability of aortic stenosis (0-100%) for each individual patient. This probability will be compared to the AI ECG result (probability 0-100%) from the patient's recently recorded 12 lead ECG which is routinely available for all patients with a recorded 12 lead ECG at our medical system.
Artificial intelligence determination of patient age by single-lead watch-based ECG | 12 months
  A previously developed AI algorithm to predict patient age from 12 lead ECG via convolutional neural network will be adapted applied to the ECGs for patients who undergo single-lead watch-based ECG recording. This neural network uses PQRST complexes to yield an ECG-predicted age. Each recorded single-lead watch-based ECG will undergo evaluation by this neural network and determine "ECG age" for each individual patient. This single-lead "ECG age" will be compared to the AI ECG "age" result determined from the patient's recently recorded 12 lead ECG which is routinely available for all patients with a recorded 12 lead ECG at our medical system.
Artificial intelligence detection of amyloidosis by single-lead watch-based ECG | 12 months
  A previously developed AI algorithm to predict potential underlying cardiac pathology assess from 12 lead ECG via convolutional neural network will be adapted applied to the ECGs for patients who undergo single-lead watch-based ECG recording. This neural network uses PQRST complexes to yield a probability of amyloidosis which may not be readily apparent via manual review. Each recorded single-lead watch-based ECG will undergo evaluation by this neural network and will produce a probability of amyloidosis (0-100%) for each individual patient. This probability will be compared to the AI ECG result (probability 0-100%) from the patient's recently recorded 12 lead ECG which is routinely available for all patients with a recorded 12 lead ECG at our medical system.

CONTACTS AND LOCATIONS:
Overall Officials: Itzhak Zachi Attia, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
Due to patient confidentiality and IRB rules, we will not make individual patient data available

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials